CLINICAL TRIAL: NCT05115344
Title: A Phase I Study Evaluating the Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Dose-escalation of Flonoltinib Maleate Tablets in Patients With Bone Marrow Proliferative Tumors
Brief Title: Study of Flonoltinib Maleate Tablets in the Treatment of Proliferative Bone Marrow Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu Zenitar Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Guizhou Bailing Group Pharmaceutical Co Ltd (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: FM-21-001
Record Dates: First submitted 2021-08-12; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Myeloproliferative Neoplasm (MPN); Myelofibrosis，MF
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- flonoltinib 25mg (Experimental): 1 case，The starting dose，Take the medicine once on D1 ，D 5 through 21.
  Interventions: Drug: flonoltinib 25mg
- flonoltinib 50mg (Experimental): 6 case，Increasing dose，Take the medicine once on D1 ，D 5 through 21.
  Interventions: Drug: flonoltinib 50mg
- flonoltinib 100mg (Experimental): 6 case，Increasing dose，Take the medicine once on D1 ，D 5 through 21.
  Interventions: Drug: flonoltinib 100mg
- flonoltinib 150mg (Experimental): 6 case，Increasing dose，Take the medicine once on D1 ，D 5 through 21.
  Interventions: Drug: flonoltinib 150mg
- flonoltinib 225mg (Experimental): 6 case，Increasing dose，Take the medicine once on D1 ，D 5 through 21.
  Interventions: Drug: flonoltinib 225mg
- flonoltinib 325mg (Experimental): 6 case，Increasing dose，Take the medicine once on D1 ，D 5 through 21.
  Interventions: Drug: flonoltinib 325mg

INTERVENTIONS:
Drug: flonoltinib 25mg — 1 case,The starting dose,Take the medicine once on D1,D 5-21.
  Arms: flonoltinib 25mg
Drug: flonoltinib 50mg — 6 case,Increasing dose,Take the medicine once on D1,D5 -21.
  Arms: flonoltinib 50mg
Drug: flonoltinib 100mg — 6 case,Increasing dose,Take the medicine once on D1,D5 -21.
  Arms: flonoltinib 100mg
Drug: flonoltinib 150mg — 6 case,Increasing dose,Take the medicine once on D1,D5 -21.
  Arms: flonoltinib 150mg
Drug: flonoltinib 225mg — 6 case,Increasing dose,Take the medicine once on D1,D5 -21.
  Arms: flonoltinib 225mg
Drug: flonoltinib 325mg — 6 case,Increasing dose,Take the medicine once on D1,D5 -21.
  Arms: flonoltinib 325mg

SUMMARY:
Flonoltinib Maleate (FM) targets Janus kinase 2 (JAK2) and FMS-like tyrosine kinase 3 (FLT3). FM is a dual target inhibitor of JAK2/FLT3.FM has the activity of inhibiting JAK2 signaling pathway, and pharmacodynamics evaluation also confirmed that FM has a good therapeutic effect on the primary splenomegaly model of mice induced by JAK2V617 mutation.Therefore, FM has the potential to treat bone marrow proliferative tumors.The drug is intended to be used in patients with MPN, mainly including medium-risk or high-risk myelofibrosis (FM) (including primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (PostPV-MF) and post-primary thrombocythemia myelofibrosis (postET-MF)), Polycythemia vera (PV) and essential thrombocythemia (ET) were the primary causes of thrombocythemia and thrombocythemia.

FM has high inhibitory activity against JAK family and FLT3 kinase, suggesting that FM may have a certain therapeutic effect on AML disease.The IC50 of JAK2 kinase inhibition by FM was as low as 0.8 nM, while the IC50 of JAK1, JAK3 and Tyk2 kinase inhibition was 690 nM, 557 nM and 65nM, respectively. The selectivity of JAK2 kinase inhibition by FM was 862.5, 696.3 and 81.3 times, respectively. Therefore, FM showed highly selective inhibition of JAK2 kinase.The IC50 for FLT3 kinase was 15 nM. FM has better inhibitory activity against JAK2 kinase than the listed Ruxolitinib and Fedratinib, and has better selectivity against JAK family.In order to determine whether FM has targets other than JAK2 and Flt3 kinases, we tested FM's inhibitory activity against 100 human kinases that are highly associated with tumors, including some common drug-resistant mutant kinases.The results showed that, except for CDK4/6, LCK and LN, FM had no obvious inhibitory activity against the screened kinases at 0.1 μm, and no other targets were found.

In vitro experiments on the proliferation of JAK2-dependent and Flt3-related tumor cell lines with FM showed that the tumor cell lines had a significant inhibitory effect. The IC50 of half of the tumor cell lines was less than 0.5 μm, which was better than or equal to the similar drugs Ruxolitinib and Fedratinib.

The effect of FM on tumor cells from MPN patients indicated that FM has the potential to treat MPN disease.

In multiple animal models of bone marrow proliferative tumors with JAK2V617F mutations, FM showed superior efficacy and low toxicity (no obvious VISCAL toxicity) than existing drugs on the market, and the tumor inhibition effect of FM showed a good dose-dependent relationship.

Objectives of Study

Main Purpose:

1. Tolerance and safety of flonoltinib maleate Tablets tablets in patients with bone marrow proliferative tumors;
2. To observe the possible dose-limiting toxicity(DLT) of flonoltinib maleate tablets in patients with bone marrow proliferative tumors,To determine the maximum tolerated dose(MTD) of flonoltinib maleate tablets,To provide the basis for the recommended dose and design scheme of the later clinical trial.

Secondary Purpose:

1. To evaluate the pharmacokinetic characteristics of single and repeated oral administration of flonoltinib maleate tablets in patients with bone marrow proliferative tumors;
2. To evaluate the primary efficacy of single and multiple oral flonoltinib maleate tablets in patients with bone marrow proliferative tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, gender unlimited;
2. Patients diagnosed as PMF, PV (PV at least 24 weeks), ET according to WHO criteria (2016 edition), or post-PV-MF or post-ET-MF according to IWG-MRT criteria;
3. Any of the following criteria is met :(1) Patients receiving treatment for myeloid fibrosis must be at least medium-risk -1 or high risk as assessed according to the DIPSS risk grouping criteria; (2) PV and ET patients who are resistant or intolerant to hydroxyurea and/or interferon therapy;
4. No immediate plans for a stem cell transplant;
5. At least 4 weeks or more than 5 half-lives (whichever is longer) after receiving the last antitumor therapy (chemotherapy, radiotherapy, biotherapy or immunotherapy) before enrollment;
6. Expected survival ≥12 weeks;
7. ECOG≤2;
8. Splenomegaly: palpate the margin of the spleen (the farthest point of the spleen) at least 5 cm below the costal margin; Or not accessible due to body type (obesity), but confirmed by MRI (CT scan if necessary) spleen assessment at screening time, the volume is ≥450 cm3;
9. Bone marrow primitive cells and peripheral blood primitive cells ≤10%;
10. PLT≥75×109 /L, ANC≥1.0×109 /μL, HGB> without the assistance of colony stimulating factor, growth factor, thrombogenic factor or platelet infusion; 80 g/L. Subjects did not receive growth factor, colony-stimulating factor, thrombogenic factor or platelet transfusions within 2 weeks before examination.
11. Heart, lung, liver, kidney, pancreas without serious organic lesions (LVEF (left ventricular ejection fraction) ≥45%; Total bilirubin ≤1.5×ULN; Serum creatinine ≤1.5×ULN or CCR> 40 ml/min. Alanine aminotransferase (ALT) ≤2×ULN; Aspartate aminotransferase (AST) ≤2×ULN;
12. No severe coagulation abnormalities (PT≤1.5×ULN, APTT≤1.5×ULN, TT≤1.5×ULN);
13. Those who agree to participate in the study and sign the informed consent;
14. Agree to comply with the regulations of the hospital and research institution.

Exclusion Criteria:

1. The toxicity of previous anticancer therapy does not recover to grade I or below (except for hair loss), or does not fully recover from previous surgery (major surgery within 4 weeks);
2. Allergic constitution, allergy to test drugs and their excipients;
3. Any significant clinical or laboratory abnormalities that the investigator considers to affect the safety reviewer, such as: A. Uncontrolled diabetes - fasting glucose > 250 mg/dL (13.9 mmol/L), b. Patients with hypertension who cannot be reduced to the following range after treatment with two or less antihypertensive drugs (systolic blood pressure < 160 mmHg, diastolic blood pressure < 100 mmHg), c. Peripheral neuropathy (NCI-CTC AE V5.0 Grade 2 or above);
4. Patients with a history of congestive heart failure, unstable angina pectoris or myocardial infarction, cerebrovascular accidents, or pulmonary embolism within the first 6 months were screened;
5. Patients with impaired heart function (Ejection fraction measured by ultrasonic electrocardiogram; ST segment descending in two or more channels in 45% or complete left bundle branch block > 1 mm or T wave inverted; Congenital ventricular arrhythmia, clinically significant tachycardia (>; 100 beats/min), bradycardia (lt; 50 times/min), ECG QTc > 450 ms (male), QTc > 480 MS (female) or clinically significant heart disease (such as unstable angina pectoris, congestive heart failure, myocardial infarction within 6 months);
6. Arrhythmic disease requiring treatment, or QTC interphase (QTCB) > 480 ms;
7. Any active infections requiring treatment at the time of screening;
8. Patients who had previously undergone splenectomy or who had received radiotherapy in the splenic region within 12 months prior to screening;
9. Positive HIV antibody, positive active hepatitis B virus (HBsAg positive, HBV-DNA positive or ≥1000 copies/mL), positive anti-HCV antibody or HCV-RNA at screening time;
10. Screening patients with epilepsy or using psychotropic drugs or sedatives;
11. Pregnant or lactating women, fertile women/men who refuse to use contraceptives during the trial and within 6 months after the trial;
12. Patients who have had malignant tumors (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) in the past 5 years;
13. Concomitant with other serious diseases that the investigator believes may affect patient safety or compliance;
14. Screening patients who participated in other new drugs or medical devices and took study drugs or used study devices within the previous 3 months;
15. Within 2 weeks before randomization and into the group to use any drug for MF (JAK inhibitor, hydroxyurea), any immune modulators (such as Sally degree amine), any immune inhibitors, 10 mg/day or prednisone or equivalent strength of biological effect of glucocorticoid, growth factors, such as EPO therapy, or within six drug half-life of patients;
16. Intravenous use of either a potent or moderate CYP3A inhibitor (such as ketoconazole, clarithromycin, itraconazole, nefazoldone, telimycin) or a potent CYP3A4 inducer (rifampicin perforatum) within two weeks prior to initial administration;
17. Patients with a history of congenital or acquired bleeding diseases;
18. Alcohol dependence or drug abuse;
19. People who use grapefruit, star fruit or its products within 48 hours before taking the study drug for the first time, or who do not agree to prohibit the consumption of the above-mentioned food, drink or other special diet, which may affect the absorption, distribution, metabolism and excretion of the study drug;
20. Other factors considered by the investigator to be unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-11-12 (Estimated); Primary Completion 2022-12-29 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Flonoltinib Maleate Pharmacokinetics (PK)：Cmax | 72hours
  Estimation of maximum observed plasma concentration
Flonoltinib Maleate Pharmacokinetics (PK)：Tmax | 72hours
  Estimation of time to reach Cmax
Flonoltinib Maleate Pharmacokinetics (PK)：AUC0-72h | 72hours
  Estimation of AUC from time zero to the last measured time point
Flonoltinib Maleate Pharmacokinetics (PK)：AUC0-∞ | 72hours
  Estimation of AUC from time zero extrapolated to infinity Estimation of AUC from time zero extrapolated to infinity Estimation of AUC from time zero extrapolated to infinity Estimation of AUC from time zero extrapolated to infinity Estimation of AUC from time zero extrapolated to infinity Estimation of AUC from time zero extrapolated to infinity
Flonoltinib Maleate Pharmacokinetics (PK)：MRT | 72hours
  Estimation of mean residence time
Flonoltinib Maleate Pharmacokinetics (PK)：Vd | 72hours
  Estimation of apparent volume of distribution
  Apparent volume of distribution
  Apparent volume of distribution
Flonoltinib Maleate Pharmacokinetics (PK)：t1/2 | 72hours
  Estimation of terminal elimination half-life
Flonoltinib Maleate Pharmacokinetics (PK)：CLz/F | 72hours
  Estimation of clearance when dosed orally
Flonoltinib Maleate Pharmacokinetics (PK)：Vz/F | 72hours
  Estimation of apparent volume of distribution when dosed orally
Flonoltinib Maleate Pharmacokinetics (PK)：Ke | 72hours
  Estimation of the elimination rate constant of a drug in the body

CONTACTS AND LOCATIONS:
Overall Officials: Lijuan Chen, doctor, Study Chair — West China Hospital

IPD SHARING:
Plan to Share IPD: No